CLINICAL TRIAL: NCT06952868
Title: A Phase II Study to Evaluate the Efficacy and Safety of the Boron Neutron Capture Therapy (BNCT) Using the B10 L-BPA as Boron Carrier in Patients With Unresectable Recurrent Head and Neck Cancers
Brief Title: Boron Neutron Capture Therapy With B10 L-BPA for Unresectable Recurrent Head and Neck Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Heron Neutron Medical Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH114-REC1-042
Record Dates: First submitted 2025-04-07; First posted 2025-05-01 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer; Boron Neutron Capture Therapy
Keywords: phase II; B10 L-BPA; BNCT
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, single-arm, Phase II clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm treated by BNCT only (Experimental)
  Interventions: Drug: Drug: B10 L-BPA Injection

INTERVENTIONS:
Drug: Drug: B10 L-BPA Injection — The investigational product is B10 L-BPA Injection, is a boron-containing compound in which 10B replaces a position on L-phenylalanine at the para position with dihydroxyboron.
  This single arm of the study is designed to evaluate the therapeutic efficacy of BNCT, wherein patients receive B10 L-BPA administration followed by neutron irradiation.

SUMMARY:
This Phase II study, titled "A Phase II Study to Evaluate the Efficacy and Safety of Boron Neutron Capture Therapy (BNCT) Using B10 L-BPA in Patients with Unresectable Recurrent Head and Neck Cancers," aims to assess the efficacy and safety of B10 L-BPA-based BNCT in this patient population. The primary objective is to evaluate its efficacy, while secondary objectives include assessing safety, survival outcomes, tumor response, and the pharmacokinetics (PK) profile of B10 L-BPA and boron.

ELIGIBILITY:
Inclusion Criteria:

1. Subject aged 18-80 (inclusive).
2. Histologically or cytologically confirmed diagnosis of head and neck cancers with no distant metastasis in subjects as follows:

   1. Unresectable recurrent or persistent squamous cell carcinoma (SCC) after completing one of the following frontline therapies:

      * Standard concurrent chemoradiotherapy with a platinum-containing regimen.
      * Curative induction chemotherapy with a platinum-containing regimen, followed by radiation therapy.
      * Radiation therapy alone in the prior treatment for those who are unfit for a platinum-containing regimen or reject chemotherapy for the treatment of locoregional recurrence.
      * Concurrent chemoradiotherapy with a cetuximab-containing regimen in the prior treatment for those who are unfit for a platinum-containing regimen or reject other chemotherapy for the treatment of locoregional recurrence.
   2. Unresectable recurrent or persistent non-squamous cell carcinoma (nSCC) after receiving any type of frontline therapies.
3. Subjects who are unsuitable for systemic therapies, or subjects who refuse systemic therapies.
4. Receipt of prior radiation therapy between 40 Gray (Gy) and 75 Gy at the target lesion(s) for SCC patients and no more than 75 Gy at the target lesion(s) for nSCC patients.
5. There must be a time interval ≥ 3 months between prior radiation therapy and the scheduled BNCT.
6. There must be a time interval ≥ 1 month between receipt of antitumor drugs and the scheduled BNCT.
7. Measurable disease by magnetic resonance imaging (MRI) and/or computed tomography (CT) scan and ≤ 7 cm in the longest dimension.
8. At least one measurable lesion that can be assessed by RECIST version 1.1.
9. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-2.
10. Life expectancy ≥ 3 months in the opinion of the investigator.
11. Adequate organ functions as defined below:

    * Hemoglobin ≥ 8.0 g/dL.
    * White blood cell (WBC) count ≥ 2.5 x 103/μL.
    * Neutrophil count ≥ 1.5 × 103/μL.
    * Platelet count ≥ 80 × 103/μL.
    * Aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal (ULN).
    * Alanine aminotransferase (ALT) ≤ 2.5 × ULN.
    * Serum creatinine ≤ 1.5 × ULN.
12. Negative serology test for human immunodeficiency virus (HIV) infection.
13. Female subject with reproductive potential must have a negative result of serum pregnancy test at the screening visit and urine pregnancy test before the B10 L-BPA administration.
14. Female subject with childbearing potential as well as male subject with reproductive potential must agree to refrain from unprotected sex and use 2 methods of highly effective contraception with their partner (e.g. barrier contraceptives [male condom, female condom, or diaphragm plus spermicide], intrauterine device, hormonal methods [hormone shot or injection, implants, combination oral contraceptives, or patches]) until the end of this study.
15. Physically and mentally capable of participating in the study and willing to adhere to study procedures.
16. Provision of signed informed consent.

Exclusion Criteria:

1. Presence of secondary cancer with the exception of carcinoma in situ and skin cancers after curative surgery.
2. Synchronous multiple head and neck cancers outside the field of neutron beam irradiation.
3. Distant metastasis outside of the head and neck region.
4. Imaging studies, e.g., CT, MRI, demonstrating tumor invasion into the carotid artery.
5. Unsuitable for the BNCT, as assessed by the investigator based on the investigator-determined computed tomography angiography (CTA) of head and neck in suspected cases of tumor invasion into the carotid artery.
6. Presence of any ≥ Grade 3 toxicity (e.g., mucositis, stomatitis, and skin inflammation) at the prior irradiation area, as assessed by the NCI-CTCAE version 5.0.
7. Presence of ≥ Grade 3 cataract, as assessed by the NCI-CTCAE version 5.0.
8. Active infections requiring systemic treatment within 2 weeks of the screening visit.
9. Myocardial infarction, unstable angina, or poorly controlled arrhythmia within 6 months prior to the scheduled BNCT.
10. Severe comorbidities including but not limited to poorly controlled epilepsy, poorly controlled diabetes mellitus, poorly controlled hypertension, chronic lung diseases, e.g., obstructive pneumonia, interstitial pneumonia, pulmonary fibrosis, and severe emphysema, kidney diseases, e.g., chronic renal failure, acute renal failure, and nephrotic syndrome, cardiac diseases, e.g., New York Heart Association (NYHA) Functional Classification Class III or IV, and/or other severe conditions in the opinion of the investigator.
11. Suspected or known hypersensitivity (including allergy) to any of B10 L-BPA components (e.g., L-phenylalanine) or contrast media.
12. History of prior BNCT.
13. Subject with hereditary fructose intolerance.
14. Subject with phenylketonuria.
15. Presence of any dental conditions necessitating tooth extraction within 2 weeks before and after the BNCT, as assessed by the dentist.
16. Restless subjects who were unable to lie or sit in a cast for more than 30 minutes.
17. Any medical or psychiatric conditions that, in the opinion of the investigator, may interfere with optimal participation in the study or place the subject at increased risk of adverse events (AEs).
18. Received any investigational drug or device or have participated in a clinical study within 4 weeks prior to the screening visit.
19. History of substance or alcohol abuse within 6 months prior to the screening visit.
20. Female subject who is planning to be pregnant or lactating during the study period.
21. Subject who is considered unfit to participate in the clinical study as assessed by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Assessment of the Efficacy of B10 L-BPA-Based BNCT in Unresectable Recurrent Head and Neck Cancers | 6 months
  The objective response rate (ORR) of the B10 L-BPA-based BNCT, as evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. ORR is defined as the proportion of subjects whose best overall response is either complete response (CR) or partial response (PR) of the target lesions.

SECONDARY OUTCOMES:
Evaluation of the Safety of B10 L-BPA-Based BNCT in Unresectable Recurrent Head and Neck Cancers | 6 months
  Safety parameters, including occurrence, severity, and relationship of the treatment-emergent adverse events (TEAEs) and adverse events of special interest (AESIs), as assessed by the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 during the study period.
Assessment of the Survival Status of B10 L-BPA-Based BNCT in Unresectable Recurrent Head and Neck Cancers | 6 months
  PFS is defined as the time from receiving the B10 L-BPA-based BNCT until progressive disease (PD) or death from any cause, whichever comes the first.
  OS is defined as the time from receiving the B10 L-BPA-based BNCT until death from any cause.
Assessment of Tumor Responses to B10 L-BPA-Based BNCT in Unresectable Recurrent Head and Neck Cancers | 6 months
  Tumor responses, including complete response (CR), partial response (PR), stable disease (SD), objective response rate (ORR), disease control rate (DCR), duration of response (DoR), time to CR, and time to PR, as evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Peak Plasma Concentration (Cmax) | 3 Days
  Maximum observed concentration of B10 L-BPA in plasma.
Time to Peak Plasma Concentration (Tmax) | 3 Days
  Time at which the maximum observed plasma concentration (Cmax) of B10 L-BPA occurs.
Area Under the Plasma Concentration-Time Curve to Last Quantifiable Concentration (AUClast) | 3 Days
  Area under the plasma concentration-time curve from time 0 to the last measurable concentration of B10 L-BPA.
Area Under the Plasma Concentration-Time Curve to Infinity (AUCinf) | 3 Days
  Area under the plasma concentration-time curve from time 0 extrapolated to infinity for B10 L-BPA.
Elimination Half-Life (t1/2) | 3 Days
  Time required for the plasma concentration of B10 L-BPA to decrease by half.
Percentage of Recovered B10 L-BPA in Urine | 3 Days
  Percentage of the administered B10 L-BPA dose recovered in urine.
Percentage of Recovered B10 L-BPA Metabolites in Urine | 3 Days
  Percentage of the administered B10 L-BPA metabolites recovered in urine.
Renal Clearance of B10 L-BPA | 3 Days
  Renal clearance rate of B10 L-BPA based on urine and plasma concentrations.

OTHER OUTCOMES:
Assessment of the Population of Circulating Immune Cells and Associated Cytokines Before and After B10 L-BPA-Based BNCT | 6 months
  Blood samples will be collected to assess MDSCs, T cells and interleukin-1 β at multiple time points: before and after BNCT. This approach aims to clarify whether the levels of circulating immune cells could serve as prognostic indicators for BNCT treatment outcomes.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - Taipei Veterans General Hsopital, Taipei,, Taipei